CLINICAL TRIAL: NCT04504292
Title: Pilot Study to Assess Tolerability and Feasibility of Oral Sulfate Solution (SUPREP) in Hospitalized Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Vanessa Shami, MD, Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 21980
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Inpatient Colonoscopy; Oral Sulfate Solution; Polyethelene Glycol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral sulfate solution (SuPREP arm) (Experimental): Per the package insert: The dose for colon cleansing requires administration of two bottles of SUPREP Bowel Prep Kit. Each bottle is administered as 16 oz of diluted SUPREP solution with an additional 1quart of water taken orally. The total volume of liquid required for colon cleansing (using two bottles) is 3 quarts (approximately 2.8 L) taken orally prior to the colonoscopy outlined below under frequency.
  Two 6 oz bottles of oral solution: Each 6 oz bottle contains: sodium sulfate 17.5 g, potassium sulfate 3.13 g, magnesium sulfate 1.6 g.
  Interventions: Drug: SUPREP Bowel Prep Kit
- Polyethelene Glycol (GoLytely arm) (Active Comparator): Polyethylene Glycol Bowel Prep Kit
  Interventions: Drug: Golytely Oral Product

INTERVENTIONS:
Drug: SUPREP Bowel Prep Kit — Bowel prep prior to colonoscopy
  Arms: Oral sulfate solution (SuPREP arm)
Drug: Golytely Oral Product — Bowel prep prior to colonoscopy
  Arms: Polyethelene Glycol (GoLytely arm)

SUMMARY:
This study will test the efficacy, tolerability, and feasibility of an oral sulfate solution (SUPREP) for inpatient colonoscopy preparation, compared to the standard of care (GoLytely). The hypothesis is that SUPREP will be well tolerated and non-inferior to standard polyethylene glycol bowel preparation for colonoscopies in an inpatient setting. To test this, at least 124 subjects who are undergoing an inpatient colonoscopy will be randomized to receive either SUPREP or standard of care. The Boston Bowel Preparation Score will be collected as standard of care for both groups. Safety will be monitored from standard of care blood tests and ECG (when indicated). Subjects will be given a survey to assess how tolerable they found the procedure.

A non-inferiority design will be used to compare SUPREP to the standard of care polyethylene glycol preparation. Data analysis will be performed on Boston Bowel Preparation Score and rate of failure of preparation (measured as number of successful subsequent colonoscopies).

ELIGIBILITY:
Inclusion Criteria:

* Patients will be approached with consent for the study only if there is a clinical indication for pursuing an inpatient colonoscopy

Exclusion Criteria:

* Inability to consent (patient or POA)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority design to compare SUPREP to GoLytely (standard of care) | 6 months
  Boston Bowel Preparation Score

SECONDARY OUTCOMES:
Failure of performing colonoscopy | 6 months
  Prep Adequacy

REFERENCES:
- [Background] Lee HH, Lim CH, Kim JS, Cho YK, Lee BI, Cho YS, Lee IS, Choi MG. Comparison Between an Oral Sulfate Solution and a 2 L of Polyethylene Glycol/Ascorbic Acid as a Split Dose Bowel Preparation for Colonoscopy. J Clin Gastroenterol. 2019 Nov/Dec;53(10):e431-e437. doi: 10.1097/MCG.0000000000001137. PMID 30308546